CLINICAL TRIAL: NCT02006355
Title: Continuous Local Anesthesia Versus Continuous Femoral Nerve Bloc After Total Knee Arthroplasty: Impact on Mean Discharge Aptitude Delay
Acronym: GLASGOW
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5560
Record Dates: First submitted 2013-11-27; First posted 2013-12-10 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous femoral nerve bloc (Active Comparator): Continuous femoral nerve bloc
  Interventions: Drug: Ropivacaine
- Continuous local anesthesia (Experimental): Continuous local infiltration of local anesthetic in the operated knee.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine

SUMMARY:
This study aims at comparing continuous local anesthesia and femoral nerve bloc for total knee arthroplasty in terms of post-operative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Total knee arthroplasty
* Age > 18 years with social security covering.
* Written informed consent

Exclusion Criteria:

* Age < 18 years
* ASA Physical Status > III
* Body weight < 50 kg
* Latex or silver allergy.
* Loco-regional anesthesia contraindication
* Chronic anticoagulant, corticoid or pain treatment.
* Rivaroxaban or enoxaparin contraindication
* Communication issues
* Patient under guardianship
* Pregnant or breast-feeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-08-12 (Actual)

PRIMARY OUTCOMES:
Discharge ability time period | Participants will be followed for the duration of hospital stay, an expected average of 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves JENNY, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- CCOM-Hôpitaux Universitaires de Strasbourg, Illkirch-Graffenstaden, France